CLINICAL TRIAL: NCT04997486
Title: The Effect of Time-restricted Eating on Liver Metabolism
Acronym: TREL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1757716
Record Dates: First submitted 2021-07-20; First posted 2021-08-09 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: NAFLD; Obesity; Nutritional and Metabolic Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Nutritional and Metabolic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Subjects will consume all meals/snacks during a ~15-h daily eating period (~9-h fasting). The prescribed energy intake will be monitored and adjusted as needed to achieve weight maintenance.
- TRE isocaloric (Experimental): Subjects will consume all meals/snacks during a ~9-h daily eating period (~15-h fasting). The prescribed energy intake will be monitored and adjusted as needed to achieve weight maintenance.
  Interventions: Behavioral: Time restricted eating
- TRE ad libitum (Experimental): Subjects will consume all meals/snacks during a ~9-h daily eating period (~15-h fasting) without any other dietary advice.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Participants will be asked consume all meals/snacks during a ~9-h daily eating period (~15-h fasting).
  Arms: TRE ad libitum; TRE isocaloric

SUMMARY:
Numerous studies have established the role of nutrition on obesity and its related metabolic diseases, which together affect a billion individuals worldwide. Evidence indicate that meal timing regulates numerous metabolic processes suggesting that meal time manipulation may be a simple intervention against obesity and its metabolic diseases. Time-restricted eating (TRE) is a dietary manipulation that involves restricting food intake to 6-10 h/day with no energy intake the rest of the day. In rodents, TRE significantly decreases hepatic steatosis and dyslipidemia, while it supports a healthier hepatic cellular content even without caloric restriction, potentially by alternating activation of nutrient sensing mechanisms and effects on circadian oscillations. However, an understanding of the effect of TRE on liver health in people is not clear. Accordingly, we will conduct a randomized controlled trial in people with overweight/obesity and hepatic steatosis to determine the effect of 9 h TRE for 12 weeks, on key metabolic outcomes in liver health: 1) intrahepatic triglyceride content using magnetic resonance imaging; 2) de novo lipogenesis during fasting and postprandial conditions using administration of deuterated water in conjunction with mathematical modeling. The proposed study will enable us to determine the effect of meal timing on metabolic function in people with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* age 25-75 years
* men and women
* body mass index 25-45 kg/m2
* clinical diagnosis of NAFLD
* self-reported habitual eating period more than or equal to 14 h per day.

Exclusion Criteria:

* shift worker, recent or expected travel crossing time zones
* fasting >12-h/day more than once a week

  *> once a week no food intake after 18:00
* habitually waking up before 04:00 and sleeping before 22:30
* unstable weight (>5% change in the last 2 months)
* diabetes mellitus or alcoholic liver disease
* sleep disorder
* history of or current eating disorder
* cancer in last 5 years
* conditions that render subject unable to complete all testing procedures
* use of medications that affect the study outcome measures or increase the risk of study procedures and that cannot be temporarily discontinued
* smoking or illegal drug use
* pregnant or breastfeeding
* having metals in the body
* cognitive impairment
* gastrointestinal or bariatric surgery that affects nutrient digestion and absorption unable to grant voluntary informed consent or comply with the study instructions individuals who are not yet adults (infants, children, teenagers)
* individuals that are unable to lie motionless on the MRI scanner for an hour or *have tattoos or tattooed eyeliner
* alcohol abuse
* prisoners

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-03-07 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Change in Intrahepatic triglyceride (IHTG) content | About 12 weeks
  IHTG will be assessed by using MRI
Change in de novo lipogenesis (DNL) | About 12 weeks
  DNL will be assessed by using administration of deuterated water and measurement of deuterium enrichment in plasma lipids
Change in glucose, free fatty acid and triglyceride levels in response to a meal | Before and after 12 weeks
  Postprandial metabolic homeostasis will be assessed by using a mixed meal tolerance test.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No